CLINICAL TRIAL: NCT03862703
Title: Feasibility and Potential Efficacy of the PTSD Help App in a Danish PTSD Population: A Randomized Controlled Feasibility Trial
Brief Title: PTSD Help - a Randomized Controlled Trial of a PTSD Mobile Health App
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: The Danish Victims Fund (Other Government)
Responsible Party: Principal Investigator, Lisa Riisager, Project manager, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MHSCRDenmarkPTSDhelp
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: PTSD; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): PTSD Help intervention combined with care as usual.
  Interventions: Device: mHealth intervention, PTSD Help app.
- Control group (No Intervention): Care as usual.

INTERVENTIONS:
Device: mHealth intervention, PTSD Help app. — Experimental group will receive the app, PTSD Help.
  Other Names: Care as usual.
  Arms: Experimental group

SUMMARY:
Due to an increase in PTSD patients seeking treatment in the Danish mental health sector and the addition of Complex PTSD to the ICD-11, there is a need to increase the effectiveness of existing treatments for PTSD. mHealth interventions have been shown to be effective in reducing PTSD symptoms with small to moderate effect sizes. Therefore, the implementation of a mHealth intervention designed for psychiatric PTSD patients as a supplement to therapy may increase treatment outcome. As no studies to date has explored the effects of mHealth interventions in the Danish mental health sector the feasibility and effect of this type of intervention needs testing.

The study's primary hypothesis is that PTSD patients in a Danish psychiatric outpatient setting will want to use a mHealth application as a supplement to care as usual (CAU). The secondary hypothesis is that PTSD patients will benefit from using a mHealth application as a supplement to CAU The study is an investigator-initiated randomized controlled feasibility trial investigating PTSD help combined with CAU compared to CAU for adults with PTSD. Eighty patients will be recruited and receive either the mHealth intervention combined with CAU or CAU alone. Primary outcome is the ratio of eligible patients that agree to participate in the study and the level of user compliance. Secondary outcome data consists of exploratory data on PTSD help on PTSD symptom severity, level of psychological distress, sleep quality, dissociation symptoms, therapy readiness, quality of life, disability levels, recovery and rumination.

This study may help increase the investigator's knowledge of possible benefits of, as well as potential barriers to, the implementation of mHealth tools. It may also provide a cost-efficient means to increase therapy outcomes and decrease the duration of suffering for PTSD patients in the Danish psychiatric sector.

DETAILED DESCRIPTION:
The primary objective for the present randomized controlled feasibility study is to assess the feasibility of using PTSD help in the MHS-CRD to inform a larger future RCT study. The secondary objective is to gather preliminary exploratory data on the effectiveness of PTSD help versus treatment as usual on a range of clinically relevant outcome variables, including exploring C-PTSD as potential moderator.

The study is an investigator-initiated randomized controlled feasibility trial investigating PTSD help combined with CAU compared to CAU for adults with PTSD. The primary outcome is the ratio of eligible patients that agree to participate in the study and do so until the end of the six-week intervention period and user compliance, that is, do the patients actively use the system after randomization, Secondary outcome data consists of exploratory data on PTSD help on PTSD symptom severity, level of psychological distress, sleep quality, dissociation symptoms, therapy readiness, quality of life, disability levels, recovery and rumination. These data will be collected on PTSD help, both as standalone intervention in the six weeks before treatment and as a supplement to treatment during the patients' psychotherapeutic treatment for PTSD. The primary outcome will be assessed continuously by logging the patient's interactions with the application. Secondary outcomes will be assessed prior to randomization and start of PTSD help intervention (week 1), at post PTSD help intervention (week 7) and at the end of psychotherapeutic treatment (week 27-29). The design of this trial has been developed using the SPIRIT 2013 guidelines (Chan et al., 2013).

Participants:

The study will recruit patients referred with PTSD symptoms to the Center for Visitation and Diagnostics (CVD) under the MHS-CRD, with the following inclusion criteria: the patient 1) must be at least 18 years old, 2) fulfil the DSM-5 PTSD diagnosis criteria, 3) be referred to PTSD care package treatment (Danske regioner, pakkeforløb for PTSD, 2017), 4) have access to a smartphone with iOS (version 10 or higher) or Android (version 5.0.1. or higher) and 5) provide informed consent. Exclusion criteria are patients with 1) suicidal risk, 2) ongoing episode of bipolar disease or psychotic disorder 3) current abuse of alcohol or drugs, 4) inability to understand and/or read Danish and 5) concurrent psychiatric or psychological treatment of PTSD outside of MHS-CRD.

Randomization:

Randomization is conducted through the data management software REDCap, which allows a setup where no one from the research team have knowledge of or access to the underlying computer-generated allocation sequence. The randomization uses permuted blocks with varying block sizes based on a computer-generated allocation sequence created by a researcher with no affiliation to the project. The randomization allocation ratio is 1:1. This procedure ensures that researchers are blind to the allocation process. The randomization procedure will be stratified by presence of Complex PTSD as measured with the International Trauma Questionnaire (Cloitre, Garvert, Brewin, Bryant, & Maercker, 2013).

Blinding:

Assessors will be blinded to the patients' group allocation during the baseline assesment, all assessment post-randomization will consist solely of self-report measures administered via email through REDCap and logging of user activity in the app. In addition, researchers will be blinded during the parts of the data analysis concerning the exploratory outcome data, but not the feasibility outcomes as the group allocation is clear from the nature of the data. Participants will be blinded during baseline assesment and unblinded after group allocation.

Procedure:

Patients referred to CVD for diagnostic screening that are diagnosed with PTSD and referred to PTSD treatment in MHS-CRD will be invited to participate in the study by the clinician conducting the screening. The invitation will include a pamphlet with information about the study and contact information for the project. If the patient gives their consent for participation, he or she will be booked for an assesment interview. Patients who provide written consent and complete the assessment interview will be randomized if the participants fulfill inclusion/exclusion criteria. Patients in the experimental group will after randomization be given immediate access to PTSD help. After three days participants will receive a phone call to ascertain whether they are experiencing any technical difficulties using the app. The second and third assessments will be administered electronically via a link to the questionnaires sent in an email through REDCap. (see figure 1 for a consort diagram)

Interventions:

PTSD help - experimental group:

The PTSD help app is designed for use in preparation for and as a supplement to psychotherapy. Its functions include: Psychoeducation about PTSD, information about PTSD treatment in Denmark, instructions in techniques for relieving anxiety (such as grounding exercises, breathing exercises, physical exercises and calming images), help towards better sleep (such as guided meditations and advice for improving sleep habits and sleep environment), options for taking personal notes on symptoms and helpful strategies that can reduce distress, tools for self-assessment and monitoring of PTSD symptoms ; (Weathers et al., 2013) and sleep quality (Sleep Condition Indicator; (Espie et al., 2014) and a crisis plan with personal contacts and contact information for psychiatric emergency services.

PTSD treatment:

All patients in the project received PTSD treatment at one of six outpatient clinics in the MHS-CRD that provides PTSD treatment. All clinics complies with official Danish recommendations for PTSD Care Packet-treatment (CP-treatment) (https://www.sundhed.dk/content/cms/91/43091_pakke-belastning-tilpasningsreaktion.pdf and https://www.regioner.dk/media/5557/pakkeforloeb-for-ptsd-voksne.pdf). PTSD CP-treatment, consists of 60 hours trauma-focused group psychotherapy or 15 hours trauma-focused individual therapy combined with other treatment elements such as assessment, psychoeducation, pharmacological counselling/treatment, social skill training, meeting with social network and monitoring. The CP includes 75 hours of treatment totally (Table 1)

Table 1:

Care package treatment for Post Traumatic Stress Disorders (PTSD) CP content PTSD Psychiatric and somatic assessment 3 h Psychometry (monitoring) and psychoeducation 2 h Group psychotherapy 60 h Psychopharmacology 2 h Social skills training and couple counselling 4 h Continuity and coherence in ongoing treatment 4 h Total 75 h

Assessment and outcome

Assessment interview:

The patient's trauma history is assessed with The Trauma History Questionaire (Green, 1996), a 24-item self-report measure of the patient's lifetime trauma history. PTSD diagnosis and comorbid disorders are assessed through the Mini International Neuropsychiatric Interview (MINI v. 7.02) (Sheenan et al., 1998), a structured diagnostic interview that assesses the presence of psychiatric disorders according to DSM-V. To ascertain whether the patient also fulfills the criteria for ICD-11 PTSD or C-PTSD, the International Trauma Questionaire is administered (ITQ) (Cloitre, Roberts, Bisson, & Brewin, 2017). ITQ is a 23-item self-report questionnaire used to distinguish between PTSD and C-PTSD as defined in ICD-11. The Personality Inventory for DSM-5 Brief Form (PID-5-BF) (Krueger, Derringer, Markon, Watson, & Skodol, 2013) and The Level of Personality Functioning Scale (LPFS-BF) (Espie et al., 2014; Hutsebaut, Feenstra, & Kamphuis, 2016) are administered to assess personality disorders. The PID-5-BF, a 25-item version, is scored on five subscales assessing the five traits that make up the maladaptive personality trait model for DSM-5, negative affect, detachment, antagonism, disinhibition and psychoticism. The LPFS-BF is a 12-item self-report questionnaire that assesses the patient's level of self- and interpersonal functioning.

Feasibility outcome:

The primary feasibility outcome is the proportion of eligible patients that participate in the study until the end. The secondary feasibility outcome is the fraction of compliant patients in the experimental group. Compliance is defined as the use of PTSD help functions (excluding self-monitoring tools) corresponding to use twice a week, assessed over 6 weeks pre-treatment and 29 weeks during the treatment period. Compliance data is collected from the tracking log of the patient's app activity through a secured webpage. In addition, compliance will be assessed through a user behaviour questionnaire, developed based on questionnaires used in earlier studies evaluating the PTSD Coach app modified for the Danish research context (Kuhn et al., 2014; Miner et al., 2016) (see appendix 2). The feasibility requirements for a future RCT will be satisfied if 50% of eligible patients agree to participate in the study and if 50% of patients in the intervention group are compliant with the use of PTSD help.

Sample size:

Due to a shortage of similar studies, it is not currently possible to conduct a calculation of optimal sample size for this study. However, as a sample size calculation is not a requirement for feasibility studies, and is in some cases even discouraged (Billingham, Whitehead, & Julious, 2013), Based on existing knowledge about feasibility study methodology (Billingham et al., 2013; Teare et al., 2014; Whitehead, Julious, Cooper, & Campbell, 2016) and a feasibility study of another mHealth tool in MHS-CRD (Fenger et al., 2016), the plan is to recruit 70 patients. With 70 patients, among which 50% are rated compliant in the primary outcome, the 95% confidence interval for proportion estimate would range between 38% and 62%, which is considered acceptable.

Results:

The primary outcome, acceptance of the randomization procedure and patient compliance is analyzed through descriptive statistics, e.g., the average usage of the system per week, as well as the proportion of patients that stay in study until the end. Analysis of between-group effects on explorative outcome measures will be analyzed with analysis of covariance, using the intervention arm as the main predictor, and baseline performance and the stratification variable from randomization as covariates. For binary outcomes (e.g., compliance), logistic will be used. Due to the exploratory nature of this feasibility study, missing data will not be imputed. Results will be presented as covariate adjusted group differences or odds ratios, along with the 95% confidence interval. If the results indicate feasibility, the investigators will proceed to a randomized controlled efficacy study.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old.
* Fulfil the DSM-5 PTSD diagnosis criteria.
* Be referred to PTSD care package treatment (Danske regioner, pakkeforløb for PTSD, 2017)
* Have access to a smartphone with iOS (version 10 or higher) or Android (version 5.0.1. or higher)
* Provide informed consent.

Exclusion Criteria:

* Suicidal risk
* Ongoing episode of bipolar disease or psychotic disorder
* Current abuse of alcohol or drugs
* Inability to understand and/or read Danish
* Concurrent psychiatric or psychological treatment of PTSD outside of MHS-CRD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Randomization ratio | 40 weeks
  Ratio of eligible patients that can be randomized
compliance with intervention | 34 weeks
  Fraction of patients that used the intervention continously until the end of the study

SECONDARY OUTCOMES:
PTSD Checklist for DSM-V | 1 month
  20 item measure measuring PTSD symptoms with scores ranging from 0-80 with higher scores indicating higher symptom severity
Dissociative Symptoms Scale | 1 week
  20 item measure measuring dissociative symptoms ranging from 0-80 with higher scores indicating higher symptom severity
the Symptom Checklist-10 | 2 weeks
  10 item measure measuring psychological distress ranging from 0-40 with higher scores indicating higher levels of distress
WHO-5 | 2 weeks
  5 item measure, measuring life quality, with scores ranging from 0-25 with higher scores indicating higher quality of life
INSPIRE | 2 weeks
  5 item measure, measuring RECOVERY, with scores ranging from 0-20 with higher scores indicating better RECOVERY
Sleep Condition Indicator | 1 month
  8 item measure measuring sleep quality with scores ranging from 0-32 where higher scores indicates better sleep quality
The University of Rhode Island Change Assessment Short version | 40 weeks
  a 16 item measure, measuring motivation for therapy, with scores ranging from 16-80
Negative Events and Results of Psychological Treatment - Revised | 40 weeks
  a 13-item measure, measuring negative effects of the intervention
the user satisfaction questionnaire | 40 weeks
  measures user satisfaction and behavior

CONTACTS AND LOCATIONS:
Overall Officials: Stine B. Moeller, Ph.D., Study Chair — Head of Research Unit
Locations (1):
- Psykoterapeutisk Center Stolpegaard, Copenhagen, Gentofte, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scharff FB, Lau ME, Riisager LHG, Moller SB, Salimi ML, Gondan M, Folke S. The PTSD help app in a Danish PTSD population: research protocol of a randomized controlled feasibility trial. Pilot Feasibility Stud. 2020 Jun 30;6:92. doi: 10.1186/s40814-020-00633-x. eCollection 2020. PMID 32617173